CLINICAL TRIAL: NCT03888183
Title: Short-term Supplemental Effect of Preservative-free Low-dose Hyaluronic Acid-containing Salt Solution on Dry Eye Disease - A Randomized, Parallel-group, Double-blind, Controlled Trial
Brief Title: Effect of Preservative-free Low-dose Hyaluronic Acid-containing Salt Solution on Dry Eye Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ing-Chou Lai, MD, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201801577A3C601
Record Dates: First submitted 2019-03-20; First posted 2019-03-25 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Dry Eye
Keywords: hyaluronic acid; salt solution; dry eye disease; ocular surface disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- salt solution without 0.15% HA (Placebo Comparator)
  Interventions: Drug: salt solution without 0.15% HA
- preservative-free 0.15% HA (Active Comparator)
  Interventions: Drug: preservative-free 0.15% HA

INTERVENTIONS:
Drug: salt solution without 0.15% HA — received AIM Artificial Tears (4 to 8 times per day) with 12 weeks
  Other Names: AIM Artificial Tears
  Arms: salt solution without 0.15% HA
Drug: preservative-free 0.15% HA — received Per-Young Eye Drops (4 to 8 times per day) with 12 weeks
  Other Names: Per-Young Eye Drops
  Arms: preservative-free 0.15% HA

SUMMARY:
This trial is a randomized, parallel-group, double-blind, controlled clinical trial to evaluate the effect of hyaluronic acid (HA) on dry eye disease.

DETAILED DESCRIPTION:
This trial is a randomized, parallel-group, double-blind, controlled clinical trial to compare intervention treatment (Per-Young Eye Drops: preservative-free 0.15% HA) against control treatment (AIM Artificial Tears: salt solution without 0.15% HA). All participants will be received Per-Young Eye Drops (4 to 8 times per day) or AIM Artificial Tears (4 to 8 times per day) with 12 weeks. Two drugs are identical in appearance and order of administration will be double-blind randomized.

Primary endpoint:

To compare the central tear meniscus height (TMHc) of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged greater than or equal to 20 years (>= 20 years).
* The symptom criterium of ocular surface disease index (OSDI) score > 13.
* One of the two following examination criteria:

  1. Central tear meniscus height (TMHc) < 0.20 mm,
  2. Noninvasive tear-break time (NITBUT) < 6 s, for at least one eye.
* Informed consent form (ICF) signed by the participant or a legal guardian.

Exclusion Criteria:

* Male or female subjects aged less than 20 years (<20 years).
* The symptom criterium of ocular surface disease index (OSDI) score < 13.
* Central tear meniscus height (TMHc) > 0.20 mm and Noninvasive tear-break time (NITBUT) > 6 s for each eye.
* Acute inflammatory eye diseases.
* Receive ocular or eyelid surgeries before 6 months (except cataract surgery).
* Allergy to HA
* Pregnancy
* Conditions judged by the investigator as unsuitable for this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-01-22 (Estimated); Study Completion 2020-03-22 (Estimated)

PRIMARY OUTCOMES:
Tear meniscus height | 4 weeks
  To compare the TMHc after blink of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA at 4 weeks.

SECONDARY OUTCOMES:
Tear meniscus height | 8 weeks and 12 weeks
  To compare the TMHc of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA .
Ocular surface disease index (OSDI) score | 8 weeks and 12 weeks
  To compare the OSDI score of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA. It was ranged from 0-100, in which higher score related to more severe symptom. It was subgroup into normal (0-12), mild (13-22), moderate(23-32), and severe (33-100).
Redness score | 8 weeks and 12 weeks
  To compare the redness score of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA. It was obtained by Keratograph® 5M, Oculus. The redness score, including total redness score, temporal and nasal bulbar scores, temporal and nasal limbal redness scores, showing the severity of dry eye. The higher redness area imply more severity of dry eye.
Lipid layer thickness | 8 weeks and 12 weeks
  To compare the lipid layer thickness of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA.
Tear film dynamics | 8 weeks, 12 weeks
  To compare the tear film dynamics of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA.
Non-invasive tear break-up time (NITBUT) | 8 weeks, 12 weeks
  To compare the NITBUT of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA.
Tear fern test | 8 weeks, 12 weeks
  To compare the tear fern test of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA.
Ocular surface staining | 8 weeks, 12 weeks
  To compare the ocular surface staining of treatment with preservative-free 0.15% HA to the treatment with salt solution without 0.15% HA. The ocular surface staining will be graded according to the Oxford Scheme. Fluorescein stain is applied on the ocular surface, and then corneal and conjunctival staining are evaluated under absorption filters. Staining will be labeled by punctate dots on a series of panels in order of increasing severity and score ranges from 0 to 5 for the treatment eye.

CONTACTS AND LOCATIONS:
Overall Officials: Ing-Chou Lai, MD, Principal Investigator — Department of Ophthalmology, Chang Gung Memorial Hospital, Kaohsiung, Taiwan
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Lemp MA, Crews LA, Bron AJ, Foulks GN, Sullivan BD. Distribution of aqueous-deficient and evaporative dry eye in a clinic-based patient cohort: a retrospective study. Cornea. 2012 May;31(5):472-8. doi: 10.1097/ICO.0b013e318225415a. PMID 22378109
- [Background] Cho WH, Lai IC, Fang PC, Chien CC, Tseng SL, Lai YH, Huang YT, Kuo MT. Meibomian Gland Performance in Glaucomatous Patients With Long-term Instillation of IOP-lowering Medications. J Glaucoma. 2018 Feb;27(2):176-183. doi: 10.1097/IJG.0000000000000841. PMID 29240600
- [Background] Ho RW, Fang PC, Chao TL, Chien CC, Kuo MT. Increase lipid tear thickness after botulinum neurotoxin A injection in patients with blepharospasm and hemifacial spasm. Sci Rep. 2018 May 30;8(1):8367. doi: 10.1038/s41598-018-26750-5. PMID 29849166
- [Background] Wang CY, Ho RW, Fang PC, Yu HJ, Chien CC, Hsiao CC, Kuo MT. The function and morphology of Meibomian glands in patients with thyroid eye disease: a preliminary study. BMC Ophthalmol. 2018 Apr 12;18(1):90. doi: 10.1186/s12886-018-0763-9. PMID 29649988